CLINICAL TRIAL: NCT04418258
Title: Evaluation of a Capillary Endoscopy Aspiration Catheter
Brief Title: Capillary Endoscopy Aspiration Catheter
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Ali Rezaie, MD, Medical Director of GI Motility Program, Cedars-Sinai Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00000319
Record Dates: First submitted 2020-05-28; First posted 2020-06-05 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Microbiota; SIBO
Keywords: Endoscopy aspiration Catheter; SIBO; Gut Microbiome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Capillary Aspiration Endoscopy Catheter group (Experimental): Small intestine aspirate suction was carried out with a capillary aspiration endoscopy catheter
  Interventions: Device: Capillary Endoscopy Aspiration Catheter
- Aspiration endoscopy catheter group (Active Comparator): Small intestine aspirate suction was carried out with an aspiration endoscopy catheter
  Interventions: Device: Endoscopy Aspiration Catheter

INTERVENTIONS:
Device: Capillary Endoscopy Aspiration Catheter — Small intestinal fluid will be suctioned with using a capillary endoscopy aspiration catheter[#CSL2182; Hobbs Medical,Inc. Connecticut, US] during upper endoscopy
  Arms: Capillary Aspiration Endoscopy Catheter group
Device: Endoscopy Aspiration Catheter — Small intestinal fluid will be suctioned with using an endoscopy aspiration catheter[#2182; Hobbs Medical,Inc. Connecticut, US] during upper endoscopy
  Arms: Aspiration endoscopy catheter group

SUMMARY:
The small intestine is an understudied frontier of microbiome research. While aspiration during endoscopy is considered the gold standard to assess small bowel bacteria, the tools for sterile retrieval are primitive and poorly validated.

Endoscopic aspiration is time-consuming and prone to contamination. Inspired by plants' ability to draw water by capillary action, a novel multi-capillary sterile system was designed which is a modified version of the conventional aspiration catheter.

The purpose of this study is to examine the time and volume capabilities of this catheter in suctioning various liquids compared to conventional aspiration catheter, in two groups, each includes 23 patients that going under endoscopy at GI lab at Cedars Sinai Medical Center. The investigator will collect up to 2 ml fluid from Duodenum- in first group by using the conventional catheter and in second group by using the capillary catheter. The time collection and the volume of samples in 2 groups will be compared.

DETAILED DESCRIPTION:
The Medically Associated Science and Technology (MAST) program at Cedars-Sinai is dedicated to the development of novel drugs and devices to diagnose and treat patients. This study designed to examine the efficiency of the aspiration capillary catheter during an endoscopy procedure. The investigators want to know if this capillary catheter can suction faster than the current commercially available endoscopic aspiration catheter.

You are being asked to take part in this research study because you are undergoing an endoscopy or esophagogastroduodenoscopy procedure as part of your clinical care.

The study will enroll up to 46 people in total. This research study is designed to test the investigational use of a modified endoscopy aspiration catheter. The original, standard endoscopy aspiration catheter has been approved by the U.S. Food and Drug Administration (FDA), but the investigational catheter used in this study, which is similar in structure, makeup, and function to this approved device, has not been approved by the FDA. During regularly conducted endoscopy procedures, investigators will use either the standard catheter or a different kind of catheter to collect up to 2 ml fluid from the small intestine. The typical catheter used for this procedure is called an endoscopic aspiration catheter. The modified catheter is a capillary aspiration catheter, which is constructed and functions a bit differently. In the lab, this capillary aspiration catheter performs more efficiently, meaning it collects the fluid faster and more successfully than the usual endoscopic aspiration catheter. The investigators hope that using this different catheter will demonstrate the same improved results when used in real situations in humans. The investigators will record how long it takes to suction a sample of the intestinal contents (2 ml, approximately two-fifths of a teaspoon). These samples will be collected solely for research purposes and will be discarded per standard after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged 18-85 undergoing esophagogastroduodenoscopy.

Exclusion Criteria:

* There are no exclusion criteria for this study as subjects will be undergoing the procedures for medical reasons and not for the purposes of this study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2020-05-20 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
The volume(millilitres) of the aspirate that will be suctioned from small intestine in two groups | 5 minutes
  The volume(millilitres) of the aspirate that collected from small intestine during upper endoscopy will be the primary end point
The time(minutes) of the aspirate collection from small intestine will be measured in two groups | 5 minutes
  The time(minutes) of the aspirate collection from small intestine will be measured in two groups

SECONDARY OUTCOMES:
The rate of adverse events such as perforation, and bleeding in two groups | 30 minutes
  The rate of adverse events at 30 minutes after endoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Ali Rezaie, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided